CLINICAL TRIAL: NCT03745859
Title: Fraxinus- Assessment of an Open Source Virtual Bronchoscopic Navigation System
Brief Title: Evaluation of a New Open Source Virtual Bronchoscope Navigation System
Status: Terminated | Type: Observational
Why Stopped: necessary upgrades of essential software were not delivered
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); SINTEF Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/302
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Bronchial Neoplasms
Keywords: Bronchoscopy; Navigation; Feasibility Studies
MeSH Terms: conditions — Bronchial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fraxinus VBN system — Open source planning tool for bronchoscopy
  Other Names: Virtual Bronchoscopic Navigation System

SUMMARY:
To evaluate the feasibility of the Fraxinus Virtual Bronchoscope Navigation (VBN) System in the bronchoscopic access to target lesions. The study emphasizes the system´s efficacy in diagnostics of peripheral pulmonary lesions and the ease of use for the operator.

DETAILED DESCRIPTION:
Multi-center study. The study explores Fraxinus which is an open source, software only, simple guiding system for bronchoscopy. The system provides 3D maps with centerline-to-target information extracted from preoperative computed tomography. The ability of the system to guide a user to a peripheral target lesion will be evaluated. During bronchoscopy any established method for diagnostic sampling is allowed. User Evaluation will be essential to decide if the Fraxinus VBN System is beneficial in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* referred to thoracic department in any of the participating hospitals with undiagnosed peripheral pulmonary lesion(s) not visible by bronchoscopy
* voluntary signed an informed consent

Exclusion Criteria:

* pregnancy
* Any patient that the Investigator feels is not appropriate for this study for any reason

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patents with undiagnosed peripheral pulmonary lesion(s) who have been recommended for bronchoscopy
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Evidence if the Fraxinus VBN System has a role in the assessment of peripheral pulmonary lesions | 48 hours
  The proportion of cases in which the use of the system is considered beneficial

SECONDARY OUTCOMES:
Diagnostic yield | 1 week
  Diagnostic success defined as cytology or biopsy with pathology
Duration of procedure | 48 hours
  Time spent with preparations and bronchoscopy
Adverse events | 48 hours
  Procedure related adverse events or unexpected incidents registrated
Operators-reported satisfaction | 48 hours
  Enquiry on main operator´s experience after end of bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Sorger, md phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided